CLINICAL TRIAL: NCT01099007
Title: Phase II: Healthy Bodies, Hearts After Menopause
Brief Title: Healthy Bodies, Healthy Hearts: A Physical Activity Intervention Trial
Acronym: HBHH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL085405; 5K23HL085405-03 (NIH)
Record Dates: First submitted 2010-04-02; First posted 2010-04-06 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Obesity; Cardiovascular Disease; High Blood Pressure
Keywords: Women; Menopause; Cardiovascular Disease; Physical Activity; Weight Loss
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Hypertension; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- At Home (Active Comparator): Participants in the At Home group receive a workbook from the research staff at their baseline visit that outlines an accepted nutrition and physical activity program to complete on their own.
  Interventions: Behavioral: At Home
- In Person (Experimental): Participants in the In Person group have weekly visits for the 12 weeks to the research office. The first visit can last up to one and a half hours and each subsequent visit can last approximately one hour. Group meetings provide appropriate nutrition and physical activity information as well as behavioral change strategies. Sessions also include some light physical activity (equal to brisk walking).
  Interventions: Behavioral: In Person

INTERVENTIONS:
Behavioral: In Person — Participants in the In Person group have weekly visits for the 12 weeks to the research office. The first visit can last up to one and a half hours and each subsequent visit can last approximately one hour. Group meetings provide appropriate nutrition and physical activity information as well as behavioral change strategies. Sessions also include some light physical activity (equal to brisk walking).
  Arms: In Person
Behavioral: At Home — Participants in the At Home group receive a workbook from the research staff at their baseline visit that outlines an accepted nutrition and physical activity program to complete on their own.
  Arms: At Home

SUMMARY:
The overall aim of Healthy Bodies, Healthy Hearts research study is to promote physical activity in women aged 45-65 years to promote reduced risk of cardiovascular disease. The investigators are conducting an intervention for 12 weeks that promotes physical activity through support groups, group exercise sessions or through information that is given at the baseline appointment. Participants will be randomly assigned to a group.

ELIGIBILITY:
Inclusion Criteria:

* Not currently exercising for at least 100 minutes per week
* Have a Body Mass Index (BMI) of 25 or greater
* Has a physician in one of the three participating practices

Exclusion Criteria:

* Not able to walk 1/2 mile or 1 flight of stairs without assistance from another person or an assistive device

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months
  The goal of the intervention is for participants to have a 10% reduction in body weight

SECONDARY OUTCOMES:
Increase physical activity | 3 months
  The goal of the study is for participants to reach and maintain an average of 150 minutes of moderate to brisk physical activity per week.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States